CLINICAL TRIAL: NCT03703843
Title: Feasibility of ARTUS MONO Artificial Urinary Sphincter Implant in Women
Brief Title: ARTUS MONO Artificial Urinary Sphincter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Myopowers Medical Technologies France SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ARTUS00
Record Dates: First submitted 2018-05-25; First posted 2018-10-12 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Urinary Incontinence,Stress
Keywords: AUS; Artificial Urinary Sphincter
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active (Experimental): ARTUS MONO
  Interventions: Device: ARTUS MONO

INTERVENTIONS:
Device: ARTUS MONO — Temporarily implant and activation of the medical device

SUMMARY:
The ARTUS MONO implant is an active implantable medical device (AIMD) that assist the urethral sphincter function of female patients suffering from moderate to severe urinary incontinence, by remotely opening and closing a cuff placed around the bladder neck. The purpose of this clinical investigation is to evaluate the feasibility of implantation of the device, its safety and its efficacy, when temporarily implanted in female patients scheduled for anterior pelvic exenteration for bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥ 18 yo
2. BMI > 18,5 and < 35
3. Patient scheduled for an anterior pelvic exenteration with ileal conduit urinary diversion
4. Signed informed consent

Exclusion Criteria:

1. Advanced bladder cancer with bladder neck and/or urethral extension
2. Past pelvic radiation therapy
3. Patient previously treated with an artificial urinary sphincter or other urogenital implant
4. Positive urine culture during the past 2 weeks
5. Indwelling bladder catheter during the past 2 weeks
6. Documented history of sensitivity to silicone
7. History of connectivitis disease
8. Immunosuppressive therapy in the last 3 months
9. Vulnerable subjects
10. Participation in any other clinical investigation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Bladder catheterization in presence of ARTUS MONO cuff | Day 0
  Injection then re-aspiration of 50 cc of saline water through 18 Fr Foley catheter

SECONDARY OUTCOMES:
ARTUS MONO cuff implant | Day 0
  Visual analogic scale (from worst to best imaginable easiness and safety)
ARTUS MONO cuff activation | Day 0
  Cuff closing to reach 10, 20 and 30% of urethral perimeter reduction

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas BARRY DELONGCHAMPS, PR, Principal Investigator — Hôpital Cochin
Locations (2):
- Thomayer hospital, Prague, Czechia
- Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided